CLINICAL TRIAL: NCT05204004
Title: A Prospective, Multicentre, Randomised, Blinded Study of Obstructive Sleep Apnoea Detection Using the Sunrise Solution
Brief Title: The Sunrise OSA Trial
Acronym: SOSAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: NHS Highlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRAS Project ID: 296444
Record Dates: First submitted 2021-06-21; First posted 2022-01-24 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: A prospective, randomised, blinded pilot study
Who Masked: Participant
Masking Description: Patients under investigation for OSA will use both devices (Sunrise solution and overnight polygraphy) simultaneously for a single overnight sleep study. They will be randomised to receive their treatment decision based on either the Sunrise solution or polygraphy. They will be unaware of which device their treatment decision was based on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunrise (Experimental): Participants under investigation for OSA will use both devices (Sunrise solution and overnight polygraphy) simultaneously for a single overnight sleep study. Participants randomised to the 'Sunrise' arm will receive their treatment decision based on the Sunrise solution.
  Interventions: Device: Sunrise
- Polygraphy (Active Comparator): Participants under investigation for OSA will use both devices (Sunrise solution and overnight polygraphy) simultaneously for a single overnight sleep study. Participants randomised to the 'polygraphy' arm will receive their treatment decision based on the polygraphy.
  Interventions: Device: Polygraphy

INTERVENTIONS:
Device: Sunrise — Sunrise (Sunrise SA, Belgium) is a novel integrated digital medicine solution for the diagnosis of OSA allowing the detection of respiratory disorders from the analysis of mandibular movements optimised by an artificial intelligence algorithm "machine learning". It is composed of a unique innovative sensor, placed on the chin during the night, connected via Bluetooth to a mobile application which guides the patients for the implementation and allows the transfer of the data collected by the sensor to a certified health host guaranteeing the security and confidentiality of medical data. The analysed data is integrated and automatically transferred into a detailed report made available to doctors via a secure website the day after the test.
  Arms: Sunrise
Device: Polygraphy — Polygraphy (Apnoealink-Air, ResMed, Australia) is a commercially available, limited-channel sleep study device which can be used in the home. Many sleep services in the UK already use the ApneaLink Air for routine screening. It is a portable device which consists of a nasal cannula to measure nasal flow and snoring, oximeter to measure pulse and blood oxygen levels, and a chest band to measure respiratory effort. It contains software which allows for the scoring of apnoeas, hypopnoea and arousals.
  Arms: Polygraphy

SUMMARY:
A prospective, randomised, blinded pilot study comparing the Sunrise solution and overnight polygraphy for the diagnosis of OSA in adult patients. Patients under investigation for OSA will use both devices simultaneously for a single overnight sleep study. They will be randomised to receive their treatment decision based on either the Sunrise solution or polygraphy. A retrospective check of their diagnosis will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18
2. Ability and willingness to provide informed consent
3. Patient referred for suspected OSA
4. BMI >28 kg/m2
5. Epworth Sleepiness Score >12
6. Reported snoring (criterion may be ignored if patient sleeps alone)
7. Patient able to use a smartphone application and having an internet connection at home

Exclusion Criteria:

1. Patient already treated for OSA
2. Patient has PSV or HGV driving license
3. Unstable cardiac disease
4. Supplemental oxygen
5. Known secondary sleep pathology e.g. Periodic Limb Movement Syndrome, Narcolepsy, Circadian Disorder, Obesity Hypoventilation Syndrome
6. Concerns about sleepy driving or any other potentially dangerous symptom from physician or urgent referral from GP when patient has been told to stop driving
7. Pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure
8. Patient whose beard is too thick to wear the Sunrise device, and who does not wish to shave
9. Patient with acrylic or painted fingernails, who does not wish to remove acrylic or paint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Time to treatment decision | From date of sleep study device dispatch until the date of treatment decision, assessed typically within 1 month but up to 6 months
  Time (days) from sleep study device dispatch to treatment decision

SECONDARY OUTCOMES:
Time to treatment decision; RBH vs NHS Scotland Sleep Service | From date of sleep study device dispatch until the date of treatment decision, assessed typically within 1 month but up to 6 months
  Time (days) from sleep study device dispatch to treatment decision; inner London (Royal Brompton hospital) vs Scottish Highlands (NHS Scotland Sleep Service)
AHI | After completion of the sleep studies and data from both devices is available; typically within 1 month but up to 6 months
  Apnoea-hypopnoea index compared between sleep study devices; Sunrise and polygraphy

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Raigmore Hospital, Inverness
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No